CLINICAL TRIAL: NCT00500669
Title: A Randomised, Blinded Study to Assess the Effect of Betadine in the Groin Wound of Patients Undergoing Primary Varicose Vein Surgery
Brief Title: A Randomised Study to Assess Betadine in the Groin Wound of Patients Undergoing Primary Varicose Vein Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitement too slow
Sponsor: Royal Hobart Hospital (Other Government)
Responsible Party: Principal Investigator, Stuart Walker, Staff Specialist vascular Surgery, Royal Hobart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H0011
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Varicose Veins; Wound Infection; Recurrence
Keywords: Varicose veins; wound infection; recurrence
MeSH Terms: conditions — Varicose Veins; Wound Infection; Recurrence | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betadine (Experimental)
  Interventions: Drug: Betadine
- Saline (Active Comparator)
  Interventions: Drug: Betadine

INTERVENTIONS:
Drug: Betadine — Topically

SUMMARY:
To investigate whether Betadine can reduce infection rates and recurrence rates following varicose veins surgery in a randomized double blind placebo controlled study.

DETAILED DESCRIPTION:
Introduction. Varicose vein surgery is common. Worldwide, the commonest indication for this type of surgery is cosmesis. However, there are also some medical indications, including venous eczema, lipodermatosclerosis and venous ulceration. The surgery is usually straight forward and can in most instances be done as a day case. Patient and medical practitioner expectations are therefore high. Surgery in the groin is notorious for its risk of wound infection. In primary varicose vein surgery, the groin wound infection can rate can be as high as 20% 1. A more realistic figure might be approximately 10% (Sains PS, Reddy KM, Jones HJS and Derodra JK. Audit of varicose vein surgery: the patients perspective. Phlebology 2005 20(4) 179 - 182.)

A small prospective study has been conducted at the Royal Hobart Hospital to establish the wound infection rate in this hospital. All procedures were performed under the care of a single surgeon who routinely soaks the groin wound in Betadine. Patients were followed up on a weekly basis for six weeks and had wound inspections by an independent nurse consultant. Of the 11 patients (five female, mean age 50.3years, range 31 - 74 years, mean weight 92kg, range 60 - 130kg, mean body mass index 41) who have now completed six weeks of follow up, there were a total of 17 groin wounds. Only one of these (6%) has had an infection. Unfortunately, this study was terminated prematurely as the independent nurse who was performing the wound assessments has been replaced and there was a lag interval of at least 6 weeks before her replacement was due to start.

One of the major problems with varicose vein surgery is the risk of recurrence. Recurrent varicose veins are more difficult to deal with than primary varicose veins and thus every effort must be made at the time of the primary surgery to perform an operation with the lowest recurrence rate. Despite adequate surgery, recurrence can develop via neovascularisation in the groin. This may be part of the normal wound healing process. If neovascularisation can be prevented, this may reduce the recurrence rate. However, this should not be at the detriment of healing of the groin wound.

Previous in vitro studies have looked at the effect of povidone-iodine on some of the components of wound healing. It can be toxic to granulocytes, monocytes and keratinocytes 2, 3 . Dilute Povidone-Iodine solutions are also known to inhibit human skin fibroblast growth in vitro 4, 5. In vivo studies, however, have failed to show any clinically significant delay in wound healing when wounds are irrigated with povidine iodine 4.

Povidine-iodine has bacteriocidal effects 6. Could it be that those groin wounds which develop an infection develop neovascularisation as part of the inflammatory response? Topical antimicrobial agents are commonly used in wound management. This is based on the premise that reduction of bacterial contamination aids wound healing. Sindelar showed that the incidence of superficial infections of surgical wounds irrigated with povidone-iodine solution prior to closure was less than wounds irrigated with saline (2.9% vs. 15.1%) 7 .

No toxicity has been reported with povidone-iodine used as a brief rinse or soak, as planned for this study.

In order to assess the effect of Betadine (10% povidone-iodine) in the groin wound on infection rates and recurrence rates in patients undergoing primary varicose vein surgery we will conduct a prospective, randomized study.

Following injury and haemostasis, hypoxia, high lactate levels and acidosis stimulate angiogenesis. Under the influence of factors such as bFGF and VEGF, endothelial cells proliferate and form capillary buds. These cells secrete matrix metalloproteases which allow vascular buds to dissect through the wound matrix while EGF and PDGF recruit pericytes which stabilise the new vessel formation (Betsholtz C, Lindblom P, Gerhardt H. Role of pericytes in vascular morphogenesis. EXS9422005; 115 - 125

Investigators. Mr. S. R. Walker - Staff Specialist, Vascular Surgery. Prof. Sinha - Associate Professor of Surgery Mr. David Cottier - Visiting Medical Officer - Vascular Surgery.

Protocol. Inclusion criteria - Patients undergoing primary saphenofemoral ligation for varicose veins (can be combined with short saphenous surgery).

Exclusion criteria - Allergy to iodine Redo groin dissections Patients having multiple avulsions only or saphenopopliteal ligation only Patients unable to return to outpatients for 6 weeks to undergo assessment with the wound care nurse

Patients admitted under the care of Prof. Sinha or Mr. S. R. Walker are to be included.

Patients suitable for the study will be recruited from the outpatient department. If the patient agrees to be included in the study, they should undergo a pre-operative venous duplex scan. This may alter the operative plan. If patients have had a duplex scan prior to a decision on surgery, this scan does not need to be repeated.

On admission for surgery the patient should undergo the usual pre-operative work up, including weight and height. Their past medical history should be recorded.

All patients should receive a pre-operative dose of low molecular weight heparin (Clexane 20mg) as thromboembolic prophylaxis. The groin area is shaved immediately before the operation. The groin and legs are prepared for surgery in the usual way using aqueous Betadine. No prophylactic antibiotics are to be given. The surgical procedure in the groin is then performed in a standard manner to expose the saphenofemoral junction. The junction and all tributaries are ligated. In all cases the long saphenous vein should be pin stripped to the level of the knee.

At this point, patients are randomized via a sealed envelope to either a saline soaked gauze or a Betadine soaked gauze placed in the groin wound. This is left in place for a minimum of one minute. Some surgeons may then chose to close the groin wound before proceeding to the avulsions while others may choose to leave the soaked swab in place while any avulsions are dealt with. The length of time the swab is left in the groin wound should be recorded.

The groin wound is then closed with vicral to the fascia and monocryl to the skin. The groin wound is dressed with a non occlusive dressing.

Post operative protocol - Patients will be booked to see the wound care consultant on a weekly basis for 6 weeks. The patients will be booked into Prof. Sinha and Mr. Walker's outpatient clinic on Thursday morning. The wound care consultant will attend these clinics to assess the wounds. The wound care consultant will be blinded as to whether saline or Betadine was used in the groin. The wounds will be classified as:

1. - normal post operative wound, no signs of infection
2. - erythema of the wound not extending for more than 5mm from wound edge
3. - erythema more than 5mm but no wound discharge
4. - discharge of pus from wound
5. - wound dehiscence with infection, presence of pus and necrotic tissue.

At the six week follow up, the patient should undergo a venous duplex scan. This scan is performed to ensure an adequate surgical procedure has been performed.

One year following the surgical procedure, patients undergo a final venous duplex scan to assess for signs or recurrence, and in particular, a recurrence in the groin.

Both post operative duplex request forms should be completed at the time of the original operation with dates on the request forms for the scans.

End points. Primary end point - groin wound infection Secondary end point - groin recurrence of varicose veins

Statistics. If use of Betadine can reduce the infection rate (from 20%) and recurrence rate by 50%, for a study with 90% power, we would require at least 100 patients in each group. This number could be more readily recruited in a multicentre study.

It is envisaged that approximate

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary saphenofemoral ligation for varicose veins (can be combined with short saphenous surgery).

Exclusion Criteria:

* Allergy to iodine
* Redo groin dissections
* Patients having multiple avulsions only or saphenopopliteal ligation only
* Patients unable to return to outpatients for 6 weeks to undergo assessment with the wound care nurse

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
groin wound infection | Up to 6 weeks post operative

SECONDARY OUTCOMES:
- groin recurrence of varicose veins | Up to one year post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Walker, MBBS, Principal Investigator — Royal Hobart Hospital
Locations (1):
- Royal Hobart Hospital, Hobart, Tasmania, Australia